CLINICAL TRIAL: NCT02203058
Title: Pursed-lips Breathing Reduces Reduces Dynamic Hyperinflation Induced by Activities of Daily Living Test in Patients With COPD
Brief Title: Pursed-lips Breathing and Dynamic Hyperinflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Prof. Dra. Anamaria Fleig Mayer, PhD, University of the State of Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PLB2014
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inspiratory capacity; Positive-pressure respiration; Exercise; Activities of daily living; COPD.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pursed-lips breathing (Experimental): All patients performed both tests (six-minute walk test and Glittre ADL test) with pursed-lips breathing.
  Interventions: Other: Pursed-lips breathing
- No pursed-lips breathing (Placebo Comparator): All patients performed both tests (six-minute walk test and Glittre ADL test) without pursed-lips breathing.
  Interventions: Other: No pursed-lips breathing

INTERVENTIONS:
Other: Pursed-lips breathing — Expiration with pursed-lips during functional capacity tests.
  Arms: Pursed-lips breathing
Other: No pursed-lips breathing — To avoid pursed-lips breathing, subjects use a a mouthpiece (2cm diameter X 2cm length) such as the one used in pulmonary functional tests.
  Arms: No pursed-lips breathing

SUMMARY:
Background: Dynamic hyperinflation (DH) is an important factor leading to dyspnea and consequent limitations in functional capacity of chronic obstructive pulmonary disease (COPD) patients. It has not been completely elucidated whether pursed-lips breathing (PLB) is able to minimize DH and its effects on exercise tolerance in these patients. The aim of this study was to evaluate the acute effect of PLB on DH and functional capacity in patients with COPD.

Design: Randomized cross-over study. Setting: The study will be conducted in an outpatient pulmonary rehabilitation program in Florianópolis, Brazil.

Subjects: Twenty-five patients with COPD (16 men, mean age 64 (7) years, FEV1=41.7 (14.7)% predicted, BMI=27.6 (5.13)kg/m2).

Interventions: Patients will randomly perform two six-minute walk tests with and without PLB (6MWTPLB and 6MWTNon-PLB) and two Glittre-ADL tests with and without PLB (TGlittrePLB and TGlittreNon-PLB).

Main measures: At baseline and immediately after the tests, the inspiratory capacity (IC) will be assessed by the slow vital capacity (SVC) maneuver.

DETAILED DESCRIPTION:
Pulmonary function testing Lung function will be tested using an Easy One spirometer (NDD Medical Technologies Inc., Zurich, Switzerland), and calibration checked before each evaluation. Spirometry will be performed in accordance with ATS/ERS standards (Miller et al, 2005). The predicted values will be calculated from the equations proposed by Pereira et al. (2007).

Inspiratory capacity (IC) measurement IC will be measured with the patient in the sitting position, using an Easy One portable spirometer (NDD Medical Technologies Inc., Zurich, Switzerland), before and immediately after the tests, by the slow vital capacity maneuver starting from a stable end-expiratory volume, in accordance with ATS/ERS standards (Miller et al,2005). A minimum of three maneuvers (maximum of eight) will be performed and, in order to be considered reproducible, two curves could not vary by more than 5% or 150mL. The higher value of two reproducible curves will be used for analysis. DH is considered when the IC decreased 10% and/or 150mL or more compared to the basal value (O'Donnell et al, 2001).

Six-minute walk test The 6MWT will be performed according to the guidelines of the American Thoracic Society (2002). Pulse oxygen saturation (SpO2; Oxi-Go, Oximeter Plus, Roslyn Heights, New York, USA) and dyspnea (Borg CR10 scale) will be measured at the beginning and at the end of the test. Predicted values for walking distance will be calculated according to Iwama et al. (2009).

Glittre-ADL test The TGlittre consists of completing a circuit as follows: from a sitting position, the subject stands up and walks along a flat 10-m long course, in the middle of which there is a two-step ladder (each step 17 cm high x 27 cm deep) to be climbed; after completing the 10 m, the subject faces a shelf containing three 1-kg objects positioned on the top shelf (shoulder height) and moves them one by one to the bottom shelf (waist height) and then to the floor; the objects are then returned to the bottom shelf and finally to the top shelf again; the subject walks back, climbing up and down the steps, until reaching the starting point (chair), sits down and immediately begins the next lap. The subjects carry a weighted backpack (2.5 kg for women, 5.0 kg for men) and are instructed to complete five laps on this circuit as quickly as possible. SpO2 and dyspnea index (Borg CR10 scale) will be measured at the beginning of the test, at the end of each lap, and at the end of the test (Skumlien et al, 2006).

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD stages 2, 3, and 4 of severity of airflow limitation
* history of smoking ≥ 20 pack-years
* clinical stability in the four weeks prior to the study protocol

Exclusion Criteria:

* long-term oxygen therapy
* current smoking
* any pulmonary disease other than COPD
* comorbidities that would compromise their ability to perform any of the evaluations in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Dynamic hyperinflation | At the beginning and immediately after de six-minute walk test and Glittre ADL test.
  Effect of pursed-lips breathing on inspiratory capacity during the six-minute walk test and Glittre-ADL test.

SECONDARY OUTCOMES:
Six-minute walk test performance | Both tests (with and without pursed-lips breathing) will be held at least two days to one week apart.
  Effect of pursed-lips breathing on the distance walked (meters) during the six-minute walk test.
Glittre-ADL test performance | Both tests (with and without pursed-lips breathing) will be held at least two days to one week apart.
  Effect of pursed-lips breathing on the time spent (minutes) performing the Glittre-ADL tes.

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria F Mayer, PhD, Study Director — Universidade do Estado de Santa Catraina
Locations (1):
- Núcleo de Aisstência, Ensino e Pesquisa em Reabilitação Pulmonar, Florianópolis, Santa Catarina, Brazil

REFERENCES:
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] O'Donnell DE, Revill SM, Webb KA. Dynamic hyperinflation and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):770-7. doi: 10.1164/ajrccm.164.5.2012122. PMID 11549531
- [Background] Iwama AM, Andrade GN, Shima P, Tanni SE, Godoy I, Dourado VZ. The six-minute walk test and body weight-walk distance product in healthy Brazilian subjects. Braz J Med Biol Res. 2009 Nov;42(11):1080-5. doi: 10.1590/s0100-879x2009005000032. Epub 2009 Oct 2. PMID 19802464
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Skumlien S, Hagelund T, Bjortuft O, Ryg MS. A field test of functional status as performance of activities of daily living in COPD patients. Respir Med. 2006 Feb;100(2):316-23. doi: 10.1016/j.rmed.2005.04.022. Epub 2005 Jun 6. PMID 15941658